CLINICAL TRIAL: NCT05208294
Title: The Role of Dopamine, Reward Learning and Prefrontal Activity in Expectation-induced Mood Enhancement
Acronym: CRC289A07
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Philipps University Marburg (Other)
Responsible Party: Principal Investigator, Erik Müller, Professor of Personality Psychology, Philipps University Marburg
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Basic Science
Other Study IDs: CRC 289 Projekt A07
Record Dates: First submitted 2021-12-21; First posted 2022-01-26 (Actual); Last update posted 2024-01-16 (Actual); Status verified 2024-01

CONDITIONS: Placebo Effect on Mood Improvement
Keywords: placebo effect; treatment expectations; depression; reinforcement learning; mesolimbic dopamine; EEG
MeSH Terms: conditions — Depression | interventions — Sulpiride

STUDY DESIGN:
Intervention Model Description: A fully crossed 2x2 placebo design will be employed by giving participants either a placebo or a sulpiride capsule in combination with a low vs. high expectation manipulation.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Participants will be blinded to the actual substance groups. In order to carry out the expectation manipulation, the clinician scientists will provide participants with substance information that is unrelated to the actual substance that is received by the participants. Hence the clinician scientists are blind to the actual substance (double blind design). Other than providing (invalid) substance information (i.e. the expectation manipulation) and drawing blood samples, the study clinicians do not take part in the remaining experimental procedure. The investigators who accompany participants throughout the experimental procedure are not aware of participants' true substance and expectation allocation.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- High expectation with sulpiride group (Experimental): Prior to the experimental procedure, participants are told by the study clinicians that an antidepressant sulpiride capsule is administrated, while participants actually receive a sulpiride 400mg-capsule (note that the dose is presumably too high to produce antidepressant effects).
  Interventions: Drug: Sulpiride 400 MG; Behavioral: High expectation manipulation
- High expectation with placebo group (Experimental): Prior to the experimental procedure, participants are told by the study clinicians that an antidepressant sulpiride capsule is administrated, while participants actually receive a placebo capsule.
  Interventions: Drug: Placebo; Behavioral: High expectation manipulation
- Low expectation with sulpiride group (Experimental): Prior to the experimental procedure, participants are told by the study clinicians that an inactive placebo capsule is administrated, while participants actually receive a sulpiride capsule (400 mg).
  Interventions: Drug: Sulpiride 400 MG; Behavioral: Low expectation manipulation
- Low expectation with placebo group (Experimental): Prior to the experimental procedure, participants are told by the study clinicians that an inactive placebo capsule is administrated, and participants actually receive a placebo capsule.
  Interventions: Drug: Placebo; Behavioral: Low expectation manipulation

INTERVENTIONS:
Drug: Sulpiride 400 MG — The substituted benzamide sulpiride is a selective D2-receptor antagonist that is generally well tolerated and has a low affinity to histaminergic, cholinergic, serotonergic, adrenergic, or GABA receptors. Sulpiride is slowly absorbed from the gastrointestinal tract and peak serum levels occur at 3 hours . In low doses (50-200 mg), sulpiride presumably blocks presynaptic autoreceptors, thereby elevating DA levels and reducing depressive symptoms, whereas higher doses lead to a predominant blockade of postsynaptic receptors. The dose in the present study (400 mg) is sufficient for behaviorally relevant modulations of dopaminergic processing with minimal risk of side effects. Note that participants in the sulpiride group actually receive a dose that is presumably too high to produce antidepressant effects.
  Arms: High expectation with sulpiride group; Low expectation with sulpiride group
Drug: Placebo — Participants receive an inactive placebo capsule.
  Arms: High expectation with placebo group; Low expectation with placebo group
Behavioral: High expectation manipulation — Participants will be told by the study clinicians that an antidepressive sulpiride capsule is administrated.
  Arms: High expectation with placebo group; High expectation with sulpiride group
Behavioral: Low expectation manipulation — Participants will be told by the study clinicians that an inactive placebo capsule is administrated.
  Arms: Low expectation with placebo group; Low expectation with sulpiride group

SUMMARY:
Although placebo effects on depressive symptoms are well documented, the underlying mechanisms and moderating factors of expectation effects on mood and depression are poorly understood. Various studies show reduced reward processing in clinical and subclinical depression, presumably due to abnormalities in the dopamine (DA) system. Here, the investigators will test whether expectation-induced mood enhancement is mediated by endogenous DA activity and reward learning, and moderated by individual differences in depression-related personality traits. Healthy participants (N=296) will be tested for potentially relevant personality traits and given an inactive substance (placebo) or a DA D2-receptor antagonist sulpiride (400 mg) in combination with a low vs. high expectation manipulation (fully crossed 2x2 placebo design) before performing a probabilistic reinforcement learning task, an effort expenditure task, and undergo a depressed mood induction procedure. Further, EEG indices will be assessed throughout the tasks.

The investigators expect that positive expectation improves participants' reinforcement learning, increases participants' willingness to make effort in order to obtain reward, and leads to less depressive symptoms as indicated by mood ratings upon depressive mood induction. If the overall effect of positive expectations is mediated by DA, high-dose sulpiride should block expectation-induced effects, i.e., the anticipated enhanced reinforcement learning and effort expenditure as well as mood improvement in the high vs. low expectation group.

DETAILED DESCRIPTION:
The placebo effect, i.e., raising expectations towards a successful treatment by applying an inactive substance, reportedly improves therapeutic outcomes in clinical trials. Although there is supporting evidence for the neurotransmitter dopamine (DA) and reinforcement learning, i.e. learning from reward and punishment, to mediate this effect, to the knowledge of the authors, no study has tested these underpinnings yet. The objective of the present project is to investigate whether expectation-induced mood enhancement is mediated by DA activity and reward learning, and moderated by individual differences in depression-related personality traits. To this end, participants will be told to either receive a placebo (low expectation) or a medicine which is labeled as antidepressant (high expectation) that improves mood. Orthogonal to this expectation manipulation, participants actually receive either 400 mg of sulpiride (sulpiride group) or a placebo (inactive substance group). Sulpiride is a selective D2-recptor antagonist which presumably elevates DA levels in low doses and has been used as an antidepressant. However, as a part of the high expectation group's expectation manipulation, while participants are told to receive an antidepressant, the sulpiride group actually receives a dose that is presumably too high to increase DA levels and produce antidepressant effects. Rather, 400mg of sulpirid presumably leads to a blockade of dopamine receptors and may thereby block expectation placebo effects. Participants then undergo three tasks, in which behavioral and computational markers of reinforcement learning and willingness to make effort in order to obtain reward are investigated. Further, mood ratings upon depressive mood induction will be assessed. In addition to participants behavioral responses, EEG indices will be recorded throughout the tasks. Prior to testing, participants will be asked to fill out questionnaires with regard to personality traits as well as reward response. In order to assess dopamine-related plasma prolactin, the study physician will draw one blood sample (ca. 8 ml) at the beginning of the testing session (at approximately 9 a.m.) and one hour after substance intake (at approximately 10 a.m.), which presumably corresponds with the latency of the peak of the prolactin response to sulpiride. Saliva and gene samples will be collected for hypotheses that are tested in the context of the overarching collaborative research center 289 and preregistered elsewhere.

It is expected that positive expectation improves participants' reinforcement learning, increases participants' willingness to make effort in order to obtain reward, and leads to less depressive symptoms as indicated by mood ratings upon depressive mood induction. If the overall effect of positive expectations is mediated by DA, high-dose sulpiride should block expectation-induced effects, i.e., the anticipated enhanced reinforcement learning and effort expenditure as well as mood improvement in the high vs. low expectation group.

Hypotheses:

1. Expectation enhancement (high vs. low) within the placebo group is associated with lower negative mood ratings after the mood induction procedure.
2. Expectation enhancement (high vs. low) within the placebo group enhances computationally modeled reward learning parameters and EEG markers of reward processing during the reinforcement learning task.
3. Within the placebo group, the expectation effect on negative mood ratings mentioned in (1) is correlated with the expectation effect on reward learning parameters in the probabilistic reinforcement learning task mentioned in (2).
4. Across the two expectation groups and within the placebo group, reward learning parameters and electrophysiological markers of reward processing are positively correlated with questionnaire measures of agentic extraversion (and negatively with self-reported depressive symptoms).
5. In the sulpiride group, the effects described in (1), (2), and (3) are lower than in the placebo group.
6. The prolactin response to sulpiride is correlated with the magnitude of expectation effects on reinforcement learning, negative mood, and self-reported agentic extraversion as well as depressive symptoms.
7. High levels of the personality trait agentic extraversion (and low levels of depressive symptoms) are associated with higher expectancy effects on negative mood.

ELIGIBILITY:
Inclusion Criteria:

* Right-handed
* Aged 18-60 years
* German native speaker
* Informed consent
* Normal or corrected sight

Exclusion Criteria:

* Current pregnancy
* Current or history of general medical, neurological or psychological disorders, which preclude sulpiride intake
* Self-reported presence of mental disorders
* Liver, kidney, and bowel disorders
* Regular smoking
* Reported alcohol abuse
* Illegal drug intake
* Regular drug intake by prescription in the past three months
* Dreadlocks
* BMI < 19 or > 30
* Unremovable metal objects around the head
* Previous knowledge of Japanese characters
* Excessive caffeine intake (> 8 cups per day)

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 297 (Actual)
Dates: Start 2021-12-09 (Actual); Primary Completion 2023-09-22 (Actual); Study Completion 2023-09-22 (Actual)

PRIMARY OUTCOMES:
The Positive and Negative Affect Schedule (PANAS) | Five time points: approximately 3 hours after treatment (i.e., substance intake), approximately 4 hours after treatment, approximately 4.5 hours after treatment, approximately 4.75 hours after treatment, and approximately 5 hours after treatment.
  With regard to depressive mood induction: the mean of participants' five mood ratings during and immediately after the mood induction procedure. Participants' current mood will be rated on a 5-point Likert scale ranging from 1 = very slightly or not at all to 5 = extremely.
The probabilistic reinforcement learning task | This will be the first task participants undergo approximately 3 hours after treatment (i.e., substance intake) followed by the two other tasks.
  With regard to probabilistic reinforcement learning: participants' reward learning rate parameter αG as estimated in computational modeling.
The Effort Expenditure for Rewards Task (EEfRT) | This will be the second task participants undergo which follows the probabilistic reinforcement learning task (approximately 4 hours after treatment) followed by the mood induction procedure.
  With regard to effort expenditure: The number of participants' choices for the hard task which required more effort.

SECONDARY OUTCOMES:
Mood ratings | Simultaneously as PANAS (see primary outcome 1).
  Several further mood items will be rated on an 8-point scale ranging from 0 = not at all to 8 = very.
EEG responses to mood induction | Approximately 4. 5 hours after treatment (i.e., during the mood induction procedure which follows the probabilistic reinforcement learning task and the EEfRT tasks).
  With regard to depressive mood: the late positive potential (LPP) in response to depressive vs. neutral statements, and frontal alpha asymmetry during the 5-minute resting phase immediately after the mood induction procedure.
EEG responses to reward feedback | Approximately 3 hours after treatment (i.e., simultaneously during the probabilistic reinforcement learning task).
  With regard to probabilistic reinforcement learning: the reward positivity and frontomedial theta power in response to positive vs. negative feedback in the task.

OTHER OUTCOMES:
State-Trait-Anxiety-Depression Inventory (STADI) | For trait aspects: one week to two days prior to the experiment; for state aspects: approximately 30 minutes before treatment.
  STADI offers separate scales for anxiety and depression and while enabling differentiation of state and trait aspects, which are rated on a 4-point scale ranging from 1 = not at all to 4 = very.
Behaviroal Approach System Sensitivity (BIS BAS) | One week to two days prior to the experiment session.
  Personality traits with regard to individual differences in reward processing are assessed ranging from 1 = totally disagree to 4 = totally agree.
Perceived Stress Scale (PSS-10) | One week to two days prior to the experiment session.
  Participants' acute stress level are assessed on a 5-point scale ranging from 0 = never to 4 = very often, with a focus on psychophysiological stress aspects.
Somatosensory Amplification Scale (SSAS) | One week to two days prior to the experiment session.
  Participants' somatosensory amplification in the development of side effects/nocebo effects are assessed on a 5-point scale ranging from 1 to 5. A higher total score indicates greater symptom amplification.
Big Five Short Screener (BFI-10) | One week to two days prior to the experiment session.
  A short scale for assessing the Big Five dimensions of personality. Statements with regard to personality are rated on a 5-point scale ranging from 1 = disagree strongly to 5 = agree strongly.
Beck Depression Inventory (BDI-II) | One week to two days prior to the experiment session.
  Self-rating scale with regard to depressiveness which is scored on a scale of 0-3 in a list of four statements arranged in increasing severity about depressive symptoms. Higher scores indicate higher degree of the presence and intensity of mood symptoms.
Generic Assessment of Side Effects (GASE) | Approximately 30 minutes prior to treatment.
  Assessment of side effects of clinical and experimental therapeutic interventions which is based on the statistics of the Food and Drug Administration, USA.
Generic Rating for Treatment Pre-Experiences, Treatment Expectations, and Treatment Effects (G-EEE) | Approximately 30 minutes prior to treatment.
  Self-report questionnaire about participants' experience, expectation and current state with regard to the treatment (i.e., sulpiride intake) are assessed on a 11-point scale ranging from 0 to 10, while higher scores indicate stronger degree of expectancy.
The Positive Valence System Scale (PVSS) | Approximately 30 minutes prior to treatment.
  Measure of response to a wide range of rewards with regard to reward-related abnormalities in depression and other disorders. Higher scores indicate stronger responding to rewards.
The Snaith-Hamilton Pleasure Scale (SHPS) | Approximately 30 minutes prior to treatment.
  Assessment of hedonic tone and its absence, i.e., anhedonia.
PANAS trait and state | For trait level, one week to two days prior to the experiment session; for state level, approximately 30 minutes prior to treatment.
  Assessment of positive and negative affect on the trait and state level, respectively.
The Temporal Experience of Pleasure Scale (TEPS) | One week to two days prior to the experiment session.
  Assessment of individual trait dispositions in both anticipatory and consummatory experiences of pleasure.
Mood and Anxiety Symptom Questionnaire (MASQ-30) | One week to two days prior to the experiment session.
  Assessment of anhedonia as well as negative affectivity.
Revised Life-Orientation-Tests (LOT-R) | One week to two days prior to the experiment session.
  Assessment of dispositional agentic extraversion and negative affectivity.
Reinforcement Sensitivity Theory Personality Questionnaire (RST-PQ) | One week to two days prior to the experiment session.
  Assessment of dispositional agentic extraversion and negative affectivity.

CONTACTS AND LOCATIONS:
Overall Officials: Erik M Mueller, Prof. Dr., Principal Investigator — Philipps University Marburg
Locations (1):
- Department of Psychology, Differential Psychology and Personality Research, Philipps-University of Marburg, Marburg, Hesse, Germany

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, SAP, Analytic Code
Time Frame: With publication